CLINICAL TRIAL: NCT04402268
Title: Efficacy of Risk Assessment for Sudden Cardiac Death in Patients With Hypertrophic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Daria Adamczak, MD, Poznan University of Medical Sciences
Other Study IDs: PoznanUMP
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: sudden cardiac death; risk assesment; HCM Risk-SCD Calculator
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low risk: Low risk of sudden cardiac death according to HCM Risk-SCD Calculator
  Interventions: Device: Cardioverter-defibrillator
- Intermediate risk: Intermediate risk of sudden cardiac death according to HCM Risk-SCD Calculator
  Interventions: Device: Cardioverter-defibrillator
- High risk: High risk of sudden cardiac death according to HCM Risk-SCD Calculator
  Interventions: Device: Cardioverter-defibrillator

INTERVENTIONS:
Device: Cardioverter-defibrillator — We analyzed how many HCM patients reached an end-point of sudden cardiac death defined as adequate intervention of cardioverter-defibrillator or sudden cardiac arrest.

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is a heart disease characterized by hypertrophy of the left ventricular myocardium and is most often caused by mutations in sarcomere genes. The structural and functional abnormalities cannot be explained by flow-limiting coronary artery disease or loading conditions. The disease affects at least 0,2% of the population worldwide and is the most common cause of sudden cardiac death (SCD) in young people and competitive athletes due to fatal ventricular arrhythmia, but in most patients, however, HCM has a benign course. Therefore, it is of utmost importance to properly evaluate patients and identify those who would benefit from a cardioverter-defibrillator (ICD) implantation.

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is a heart disease characterized by hypertrophy of the left ventricular myocardium and is most often caused by mutations in sarcomere genes. The structural and functional abnormalities cannot be explained by flow-limiting coronary artery disease or loading conditions. The disease affects at least 0,2% of the population worldwide and is the most common cause of sudden cardiac death (SCD) in young people and competitive athletes due to fatal ventricular arrhythmia, but in most patients, however, HCM has a benign course. Therefore, it is of utmost importance to properly evaluate patients and identify those who would benefit from a cardioverter-defibrillator (ICD) implantation.

This study assesses the accuracy of the HCM SCD-Risk Calculator, recommended by European Society of Cardiology guidelines, in patients treated in the Ist Department of Cardiology of Poznan University of Medical Sciences from 2005 to 2018.

The study group consisted of 252 patients aged 20-88 (mean 53,8 ± 15,1, median 54); 49,6% were men. The protocol consisted of medical history collection (including a questionnaire), physical examination and additional tests such as echocardiography with the assessment of global longitudinal strain and average strain, cardiac magnetic resonance, ambulatory ECG monitoring, control of implantable devices and exercise testing.

ELIGIBILITY:
Inclusion Criteria:

1. Hypertrophic cardiomyopathy,
2. Minimum 18 years,
3. Questionnaire,
4. Assessment of HCM SCD-Risk Calculator at the beginning of the observation,
5. Regular visits in Cardiology Outpatient Clinic,
6. Agreement to participate in the study

Exclusion Criteria:

1. Poorly controlled hypertension (systolic pressure on the next two visits in the Cardiology Outpatient Clinic >180 mmHg),
2. Haemodynamically significant valvular heart disease or valve replacement condition,
3. Past myocardial infarction (haemodynamically significant changes found in coronarography),
4. Heart transplant,
5. Insufficient amount of data from the subject and additional tests allowing for further analysis,
6. Lack of consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group consisted of 252 patients with hypertrophic cardiomyopathy aged 20-88 (mean 53,8 ± 15,1, median 54); 49,6% were men.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Sudden cardiac death (SCD) in risk groups | 2005-2018
  Number of SCD cases in each of risk groups according to HCM Risk-SCD Calculator

SECONDARY OUTCOMES:
New risk factors of sudden cardiac death (SCD) | 2005-2018
  New echocardiographic features, such as glibal longitudinal strain, average strain, left atrial volume index, which allow to better estimate the risk of SCD

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan Univeristy of Medical Sciences, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No
Not possible due to Polish law regulations.